CLINICAL TRIAL: NCT03981913
Title: Study of the Neuronal Substrates of the Cognitive Action Control in Parkinson's Disease Using High Density EEG
Brief Title: Cognitive Control in Parkinson's Disease
Acronym: EEGControl
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Université de Rennes, Laboratoire du Traitement du Signal et de l'Image (LTSI) (Unknown); Institut des Neurosciences Cliniques de Rennes (INCR) (Unknown); Association des Parkinsoniens d'Ille-et-Vilaine (APIV) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 35RC19_8963_EEGControl; 2019-A00608-49 (Other: ANSM ( french national agency for drugs))
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Parkinson's Disease
Keywords: Cognitive action control; Parkinson's disease; high-density EEG; theta oscillations; medial frontal cortex
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control (HC): Participants without neurological or psychiatric disturbance (n= 30)
  Interventions: Behavioral: Simon Task with high-density EEG recording
- Parkinson's disease (PD): Participants with idiopathic Parkinson's disease but without other neurological or psychiatric disturbance (n= 30)
  Interventions: Behavioral: Simon Task with high-density EEG recording

INTERVENTIONS:
Behavioral: Simon Task with high-density EEG recording — The scalp electrical activity will be collected by a 256-electrodes EEG montage (Electrical Geodesics Inc).
  During the task, participants will be asked to answer on a right or left button according to the color of a circle (yellow or blue) presented on the left or right side of a screen. Participants will have to ignore the stimulus position and respond only according to its color. This leads to two experimental conditions When the color of the circle and its position indicate the same answer, the situation is congruent and the answer is facilitated. Conversely, when they indicate two opposite responses, a conflict between the two alternative actions appears and must be resolved to provide a correct answer. This situation is said to be incongruent. At each trial, the stimulus is shown to the left or right of a central fixation cross. The participants then have to answer on a right or left button. At each trial, the reaction time and the accuracy of the response will be collected.

SUMMARY:
Cognitive action control allows resisting to irrelevant information to easily produce desired goal-directed behaviors. This cognitive process is disturbed in patients with Parkinson's disease (PD). However, the neural signature of this impairment has not been clarified yet. Several studies using electroencéphalography (EEG) showed that conflict situations in healthy participants are inevitably associated with a power increase of neuronal oscillations in the theta frequency band (~4-8Hz) in the medial frontal cortex (MFC). Conflict situations are also associated with theta functional connectivity between the MFC and task-relevant brain areas. The theta power increase and connectivity are respectively interpreted as a marker of the integration of conflicting information and as a candidate for communication between the brain areas involved in implementing cognitive action control. The objective of this project is to test the hypothesis that the deficit of cognitive action control observed in PD comes from a lack of integration of the conflict information and / or communication of this information between the MFC and other task-relevant brain areas. Investigators willl study this cognitive process using a classic conflict task, the Simon task, and by recording brain activity using high density EEG coupled with cortical source connectivity analyses. The results will allow us to evaluate whether theta oscillations can serve as a marker of cognitive control disorders in Parkinson's disease.

DETAILED DESCRIPTION:
Alterations in cognitive action control in patients with PD are well described from a behavioral point of view. However, there is currently very little information to directly link these difficulties to functional alterations of brain areas, or of efficient communication within large scale brain networks. Thus, the objective of this project is to specify the neuronal substrates linked to the difficulties in cognitive action control observed in patients with PD. The rational is based on the recent findings on the role of theta (4-8 Hz) neuronal oscillations in cognitive action control. Indeed, converging evidence linked this process to an increase in theta oscillatory power around midfrontal electrodes (FCz, Cz) and to an increase in theta functional connectivity with task-relevant brain areas.

The working hypotheses are based on the hypothesis proposed by Cohen (2014). It proposes that the medial frontal cortex (MFC; around the pre-SMA) would be involved in the integration of conflicting information, observable by studying theta oscillations' power. On the other hand, the phase synchronization of theta oscillations between the MFC and the other task-relevant cortical areas would reflect the degree of recruitment of the entire network participating in the implementation of an efficient cognitive control. Thus, according to this model, a conflict situation would lead to two main measurable electrophysiological reactions in the cortex: i) an increase in the power of theta oscillations around the MFC, ii) an increase in theta phase synchronization between the MFC and the other cortical areas (such as the lateral prefrontal and parietal cortices) involved in implementing cognitive action control. These two electrophysiological effects will be the main judgment criteria of this study.

The hypothesis is that the behavioral difficulties in cognitive action control observed in PD patients stem from a lack of integration of the conflicting information and / or a weaker communication of this information to the areas implementing the cognitive control of the action. The alteration of one or both of these aspects may explain the weaker cognitive action control observed in patients. Moreover, by inspecting the disrupted brain networks, it will be able to make hypotheses explaining the alteration of cognitive control in PD. For example, a weaker functional connectivity between the MFC and the posterior parietal cortex could indicate a lower redirection of attentional resources following the presentation of a conflictual stimulus. Another possibility would be a weaker functional connectivity between the MFC and the inferior prefrontal cortex, which would rather indicate a lack of recruitment of the inhibitory system.

The main hypothesis will be tested by comparing the performance of a group of PD patients to that of a group of healthy participants whose brain activity will be collected during the realization of a Simon task via a high resolution electroencephalography system. The behavioral performances will be compared as well as the source-reconstructed electrophysiological data. Specifically, the power of the theta oscillations within the medial frontal cortex, as well as the phase synchronization between the other cortical areas involved will be compared between the two groups. Brain-behavior relationships will also be investigated in order to try to link PD behavioral impairments to changes in theta oscillatory power/connectivity.

ELIGIBILITY:
Inclusion Criteria:

Applicable to all participants (HC and PD patients):

* Age over 18
* Correct or corrected-to-normal vision
* Affiliation to a social security scheme
* Subject having received the information on the protocol and having not manifested his/her opposition to participate.

Exclusive to patients:

- Idiopathic Parkinson's disease according to the criteria of the United Kingdom Parkinson's Disease Brain Bank Society

Exclusion Criteria:

Applicable to all participants (HC and PD patients):

* Inability to understand the information given about the study or to perform the experimental task;
* Major cognitive impairment (Moca<22) or severe neurocognitive disorder according to the DSM-V (Diagnostic and statistical manual of mental disorders -V);
* Motor difficulties preventing the performance of the task
* Addiction to drugs or alcohol;
* Major person subject to legal protection (safeguard of justice, guardianship), persons deprived of their liberty.
* Present or past moderate to severe psychiatric pathology (obsessive-compulsive disorder, bipolar disorder, schizophrenia, etc.);

Exclusive to patients:

* Present or past neurological pathology other than Parkinson's disease (cerebrovascular accident, head trauma, etc.);
* Treatment by deep brain stimulation.

Exclusive to healthy participants:

- Present or past neurological pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PD patients will be recruited from the Neurology unit of the Rennes University Hospital. The study will be proposed to them during their hospitalization, which is independent from this study and occurs as part of their routine care. Most patients are hospitalized in order to conduct pre-surgical evaluations before deep brain stimulation. No changes in treatments or any other type of routine care will be made during this study.
  HC volunteers will be recruited from the general population using a volunteer database from our lab. HC's travel expenses will be refunded by the hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Difference in theta source connectivity between PD patients and matched HC in the medial-frontal-prefrontal-parietal regions following conflict situations | 45 minutes
  The scalp electrical activity will be collected by a 256-electrodes EEG montage (Electrical Geodesics Inc.) placed in the 10-20 and 10-5 systems with a 1000 Hertz sampling rate. The 256 electrodes are arranged on a cap, the electrode placement takes only 5 minutes. Before applying the cap, we will have measured the cranial perimeter of the participant to choose the most suitable cap, three sizes of caps being available. A baseline period will be obtained by recording a 10 minutes resting state activity.

SECONDARY OUTCOMES:
Difference in MFC theta source power between PD patients and matched HC following conflict situations | 45 minutes
  The scalp electrical activity will be collected by a 256-electrodes EEG montage (Electrical Geodesics Inc.) placed in the 10-20 and 10-5 systems with a 1000 Hertz sampling rate. The 256 electrodes are arranged on a cap, the electrode placement takes only 5 minutes. Before applying the cap, we will have measured the cranial perimeter of the participant to choose the most suitable cap, three sizes of caps being available. A baseline period will be obtained by recording a 10 minutes resting state activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Houvenaghel, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided